CLINICAL TRIAL: NCT06788054
Title: Effect of a 12-week Intradialysis Exercise Program on Functional Capacity, Body Composition and Survival in Hemodialysis Patients: a Randomized Clinical Trial
Brief Title: Intradialysis Exercise Functional Capacity, Body Composition and Survival in Hemodialysis Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Martha Jocelyne Piñon Ruiz, principal researcher, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CEPIUG-P59-2024
Record Dates: First submitted 2025-01-03; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Hemodialysis; Kidney Disease, Chronic; Physical Activity; Physical Deconditioning; Physical Function; Survival; Body Composition
Keywords: hemodialysis; physical capacity; chronic kidney disease; body composition; intradialysis exercise
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study studied in hemodialysis patients the impact of intradialysis exercise on body composition, physical capacity and survival.
  This clinical trial will be carried out based on the design of groups of HD patients assigned in a randomized manner; The intervention group will receive an intradialysis aerobic exercise and muscular endurance program during the second hour of dialysis, with a frequency of three times a week during; The second group (control group) will not receive intradialytic exercise, although they will receive guidance to carry out a standard treatment, in which they will be recommended to perform aerobic and muscular resistance exercise in their homes at a frequency of three times a week, for 12 weeks .
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients with chronic kidney disease on hemodialysis with intradialytic exercise (Experimental)
  Interventions: Other: intradialysis exercise
- patients with chronic kidney disease on hemodialysis without intradialytic exercise (No Intervention)

INTERVENTIONS:
Other: intradialysis exercise — moderate intensity aerobic and muscular resistance exercise protocol lasting 12 weeks
  Arms: patients with chronic kidney disease on hemodialysis with intradialytic exercise

SUMMARY:
Chronic kidney disease and renal replacement treatments (hemodialysis, peritoneal dialysis, kidney transplant) produce various alterations at the level of muscle, bones, fat content and the heart; can alter physical capabilities such as muscle strength, resistance to climb a step repeatedly intensely, and the ability to move the joints freely, in addition to producing an increase or decrease in weight and alterations in its distribution (for example, decreasing muscle and increase fat). The above, added to the particular factors of hemodialysis such as the reduction in daily time to exercise due to the sessions, or the fatigue after it, can together generate greater repercussions on functional capacity and thus increase the risk of suffering from cardiovascular problems. and accelerate the evolution of the disease.

Therefore, this study aims to determine the effect of a 12-week supervised physical exercise program during hemodialysis on strength and ability to move, the amount of fat and muscle in the body, as well as bone wear. ; and compare these results with a group of patients who do not perform supervised exercise. In addition, it will be determined how exercise can act in the long term, preventing the risk of hospitalization and death due to cardiovascular causes. The above is useful in order to establish recommendations and protocols that help us increase the quality of life and survival of the person.

DETAILED DESCRIPTION:
Background: In Mexico, Chronic Kidney Disease (CKD) has a high prevalence and is considered one of the leading causes of death. Hemodialysis (HD) is the primary renal replacement therapy; however, it is associated with significant declines in functional capacity, body composition alterations, morbidity, hospitalization, and mortality with rates that can be 30% higher than those in the general population not on HD. It is estimated that 50% of patients die within the first three years of starting HD, primarily due to cardiovascular complications. Intradialytic exercise has been linked to improvements in functional capacity and metabolic and cardiovascular parameters in HD patients. Despite these benefits, there are few studies examining the relationship between intradialytic physical exercise and increased survival in CKD patients.Objective: To analyze the effects of a 12-week intradialytic exercise program on functional capacity, body composition, and survival in patients undergoing hemodialysis. Hypothesis: A 12-week intradialytic exercise program will improve functional capacity, body composition, and survival rates in hemodialysis patients. Materials and Methods: This clinical trial will utilize a randomized design with two groups of HD patients. The intervention group will participate in an aerobic and muscular resistance exercise program during the second hour of dialysis, three times a week for 12 weeks. The control group will not participate in intradialytic exercise but will receive guidance on standard treatment, including recommendations for aerobic and resistance exercises at home three times a week. All participants (both the intervention and control groups) will be assessed for body composition using bioelectrical impedance analysis, functional capacity through the 6-minute walk test, the 30-second sit-to-stand test, and muscle strength measured by hand dynamometry. The primary outcome variable will be the survival rate at eight months of follow-up after the exercise intervention, and during this time, the International Physical Activity Questionnaire (IPAQ-short version) will be administered every two months.

ELIGIBILITY:
Inclusion criteria:

1. Male and female patients aged between 18-50 years.
2. Patients who receive regular hemodialysis sessions 3 times a week, reported through the clinical record.
3. Patients with a clinical history of being treated with HD for at least 1 previous year (reported by clinical record).
4. Patients without a history of myocardial infarction in the last 3 months (reported by clinical record).
5. Patients who are not in a kidney transplant protocol to be performed during the next 12 months.
6. Patients who have permission from their nephrology specialist to participate.
7. Patients who agree to participate in the study, and who voluntarily sign the informed consent (IC) form.
8. Patients without a history of coronary artery disease in the last 4 months (reported by clinical record).
9. Patients without myocardial instability (angina, decompensated congestive heart failure, severe arteriovenous stenosis, uncontrolled arrhythmias), reported by clinical record.
10. Patients without active infectious process (reported by clinical record).
11. Patients without extreme changes in blood glucose levels (hyperglycemia or hypoglycemia), reported by clinical record.
12. Patients without neurological, respiratory or skeletal muscle diseases or disorders that are aggravated by exercise (reported by clinical record).
13. Patients without inability to sit, stand or walk without assistance (walking device such as cane or walker is allowed) self-reported.
14. Patients without severe anemia (Hb < 8.0 g/dL), reported by clinical record.
15. Female patients should not be under sex hormone treatment or hormone replacement therapy for menopause (self-reported).
16. Patients without lupus erythematosus as the etiology of CKD, reported by clinical record.
17. Physically inactive (Do not perform physical exercise of more than 150 minutes per week on a regular basis according to data from the World Health Organization).
18. Patients who do not have amputations of any of the extremities.

Exclusion criteria:

1. If the patient presents any disease, or neurological, respiratory or skeletal muscle disorder during the development of the physical capacity tests, or during the execution of the protocol, which is aggravated by the practice of physical exercise.
2. When the patient voluntarily decides to leave the study.
3. When the patient begins additional strength or aerobic training.
4. Patients who receive a kidney transplant during the development of the exercise protocol or follow-up during the 8-month follow-up period.
5. Patients who decide to belong to the group that will perform intradialytic exercise.
6. When for any reason the exercise is suspended for more than three continuous times.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Handgrip strength | This test will be measured before starting the intervention with intradialysis exercise and 12 weeks after the start of the same.
  Handgrip strength will be assessed with a dynamometer, which is measured in kilograms (kg). This will be measured on a day without dialysis from the arm without an arteriovenous fistula for patients with a fistula and the dominant hand for patients with a central venous catheter. The test will be performed according to the instructions of the American Society of Hand Therapists, the patient will exert the greatest possible grip strength by flexing the fingers of the hand to the maximum.Three evaluations will be carried out, considering a one-minute rest between each one, and the one in which the patient manages to exert the greatest grip will be taken into account.
Cardiorespiratory capacity | This test will be measured before starting the intervention with intradialysis exercise and 12 weeks after the start of the same.
  Cardiorespiratory capacit will be assessed using the 6-minute walk test, which is measured in meters walked. It is a validated assessment tool for exercise capacity in hemodialysis patients. The test will be performed in a hallway 30 meters long, with a flat surface. During the test, the hallway must be free of any other person's traffic. The hallway will have marks at the start and end of the route, and a mark will be placed every three meters to make the count more accurate. In addition, cones will be placed 0.5 meters after the start and 0.5 meters before the end of the route, which will serve as a reference for the participant to make the turn. All participants will be instructed to make as many laps as possible around the hallway, at the highest speed, but always safely (without running). The meters walked (estimated by the number of laps made) by the patient during the 6 minutes will be counted.
Lower limb functionality: | This test will be measured before starting the intervention with intradialysis exercise and 12 weeks after the start of the same.
  It will be evaluated by the 30-Sit to stand test through the number of times the patient "gets up and sits" in the chair for 30 seconds, it is a useful, inexpensive, portable and easy to administer test to assess the strength and functional performance of the lower extremities. A 45 cm high and 61 cm deep steel chair will be placed against the wall and the patient will be positioned sitting in the middle of the chair with his back straight, feet flat on the floor and arms crossed on the chest without leaning on the chair, from this position and at the signal "attention - now" the participant will get up completely and return to the initial position as many times as possible during 30 seconds.
Body Weight | This test will be measured before starting the intervention with intradialysis exercise and 12 weeks after the start of the same.
  body weight (kilograms) will be assessed using a Tanita brand scale, model HD-366.
Height | This test will be measured before starting the intervention with intradialysis exercise and 12 weeks after the start of the same.
  Height (centimeters) will be evaluated a Seca brand stadiometer, model 213.
Waist circumference | This test will be measured before starting the intervention with intradialysis exercise and 12 weeks after the start of the same.
  Waist circumference (centimeters) with a non-deformable measuring tape (Lufkin W606PM).
Body Mass Index | This test will be measured before starting the intervention with intradialysis exercise and 12 weeks after the start of the same.
  Body mass index (BMI) (kg/m²) will be evaluated dividing the weight in kilograms by the square of the height in meters (BMI = weight [kg]/height [m²]).
Body composition | This test will be measured before starting the intervention with intradialysis exercise and 12 weeks after the start of the same.
  For the evaluation of body composition, the bioelectrical impedance technique will be used using the Inbody brand equipment, model S10. With this equipment, the following parameters will be evaluated: percentage and content of fat mass (grams), fat-free mass (grams), visceral fat area (cm), skeletal muscle mass (grams), total body water (liters).
  The evaluation will be carried out 30 minutes after the end of the hemodialysis session, on a dialysis day because it is necessary to avoid as much as possible the excess of body water on the day of the evaluation.

SECONDARY OUTCOMES:
Metabolic variables | This test will be measured before starting the intervention with intradialysis exercise and 12 weeks after the start of the same.
  Will be evaluated of serum levels of hemoglobin (g/dL), creatinine (mg/dL), urea (mg/dL), albumin (g/dL), sodium (mEq/L), potassium (mEq/L) and calcium (mg/dL) will be determined in participants in both groups.
  Laboratory analyses will be performed on a day when patients (in the intervention and control groups) are not attending the dialysis procedure and under fasting conditions of at least 8 hours, on any of the three days prior to the start of the exercise sessions. This procedure will be repeated within the three days following the end of the exercise protocol. The control group will be evaluated at the same times as the intervention group.

CONTACTS AND LOCATIONS:
Locations (1):
- Departamento de Ciencias Médicas Universidad de Guanajuato, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: Start: January 20, 2025. End May 30, 2026